CLINICAL TRIAL: NCT03355443
Title: Efficacy of Segmental Re-examination and Retroflexion of Proximal Colon for Adenoma Miss Rate During Colonoscopy
Brief Title: Examining Techniques on Adenoma Miss Rate in Proximal Colon
Acronym: SINOCOLO2017
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, En-Da Yu, Director of Department of Colorectal Surgery and Vice Director of GI Endoscopy, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SINOCOLO2017; 2017YFC1308802 (Other Grant/Funding Number: National Key R&D Program of China)
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Colorectal Adenoma; Colorectal Polyp
Keywords: Colonoscopy; Lower Gastrointestinal Tract; Re-examination; Retroflexion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Re-examination Group (Active Comparator): Routine intubation is performed. After cecal intubation, the cecum and ascending colon is examined with colonoscope tip in forward direction for the first time. Re-intubation is performed after the first examination of the cecum and ascending colon, and then this region of the large bowel is re-examined in the same fashion. After that, the rest of the colon is examined in routine method.
  Interventions: Procedure: Re-examination
- Retroflexion Group (Experimental): Routine intubation is performed. After cecal intubation, the cecum and ascending colon is examined with colonoscope tip in forward direction for the first time. Re-intubation is performed after the first examination of the cecum and ascending colon, and then this region of the large bowel is re-examined with the colonoscope tip in reverse direction (retroflexion fashion). After that, the rest of the colon is examined in routine method.
  Interventions: Procedure: Retroflexion

INTERVENTIONS:
Procedure: Retroflexion — Retroflexion technique in colonoscopy means turning the colonoscope tip 180 degree in order to look backward in the colon and rectum.
  Arms: Retroflexion Group
Procedure: Re-examination — Re-examination in colonoscopy means examining the cecum and ascending colon twice in the routine fashion.
  Arms: Re-examination Group

SUMMARY:
The primary aim of this study is

- to explore the usefulness of re-examination and retroflexion on adenoma miss rate (AMR) in the proximal colon.

Other aims include to explore the data below when re-examination or retroflexion is used.

* Adenoma detection rate, ADR
* Polyp miss rate, PMR
* Polyp detection rate, PDR
* Withdrawal time, WT

DETAILED DESCRIPTION:
AMR = number of adenomas missing during the first examination/ total number of adenomas in both examinations = number of adenomas detected only in the second examination/(number of adenomas detected during the first examination + number of adenomas detected only in the second examination)

ELIGIBILITY:
Inclusion Criteria:

* Patients between 45 and 80 years who undergo colonoscopy examination for screening, and who receive primary screening and get positive result

Exclusion Criteria:

* Pregnant female patients
* Patients received colonoscopy in the past 5 years
* Patients who have history of colorectal cancer, colorectal polyposis, inflammatory bowel disease or heredity colorectal neoplasm syndrome such as familiar adenomatous polyposis, Lynch Syndrome and so on
* Patients who had previous abdominal surgery
* Patients who are known to have colonic stricture or obstructing tumor from the results of radiography (X ray, CT scan or barium enema)
* Patients who are presenting acute surgical conditions such as severe colitis, megacolon and active gastrointestinal bleeding
* Patients who have inadequate bowel preparation
* Patients who reject to participate in this study

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adenoma miss rate in the proximal colon (AMR) | At the end of the procedure, up to 1 hour
  AMR refers to the rate of adenoma missing, calculated as the proportion of adenomas which are missing in the first examination. AMR in the proximal colon is calculated with only the proximal colon concerned.

SECONDARY OUTCOMES:
Adenoma Detection Rate in the proximal colon (ADR) | At the end of the procedure, up to 1 hour
  ADR refers to the rate of adenoma detection, calculated as the proportion of subjects with at least one adenoma. ADR in the proximal colon is calculated with only the proximal colon concerned.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - the Sixth affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhongshan Hospital affiliated to Fudan University, Shanghai
  - Tianjin Renmin Hospital, Tianjin

REFERENCES:
- [Result] Kushnir VM, Oh YS, Hollander T, Chen CH, Sayuk GS, Davidson N, Mullady D, Murad FM, Sharabash NM, Ruettgers E, Dassopoulos T, Easler JJ, Gyawali CP, Edmundowicz SA, Early DS. Impact of retroflexion vs. second forward view examination of the right colon on adenoma detection: a comparison study. Am J Gastroenterol. 2015 Mar;110(3):415-22. doi: 10.1038/ajg.2015.21. Epub 2015 Mar 3. PMID 25732415
- [Result] Lee HS, Jeon SW, Park HY, Yeo SJ. Improved detection of right colon adenomas with additional retroflexion following two forward-view examinations: a prospective study. Endoscopy. 2017 Apr;49(4):334-341. doi: 10.1055/s-0042-119401. Epub 2016 Dec 8. PMID 27931050
- [Result] Hewett DG, Rex DK. Miss rate of right-sided colon examination during colonoscopy defined by retroflexion: an observational study. Gastrointest Endosc. 2011 Aug;74(2):246-52. doi: 10.1016/j.gie.2011.04.005. Epub 2011 Jun 15. PMID 21679946
- [Derived] Wang CL, Zhao ZY, Wu JY, Yan FH, Yuan J, Xing JJ, Wang H, Yu ED. Efficacy of cecal retroflexion observed on adenoma missing of ascending colon during colonoscopy: A prospective, randomized, pilot trial. Medicine (Baltimore). 2023 Aug 25;102(34):e34806. doi: 10.1097/MD.0000000000034806. PMID 37653767